CLINICAL TRIAL: NCT02949661
Title: Local Wound Infiltration Versus Bilateral Superficial Cervical Plexus Block With Levobupivacaine for Upper Tracheal Resection and Reconstruction Surgery Under General Anesthesia.
Brief Title: Local Wound Infiltration for Tracheal Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of interest in the subject
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: R ∕16.08.18
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Upper Tracheal Resection; Tracheal Reconstruction Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Superficial cervical plexus block (Experimental): Patients will receive bilateral superficial cervical plexus block using levobupivacaine
  Interventions: Procedure: Superficial cervical plexus block
- Local wound infiltration (Active Comparator): Patients will receive local wound infiltration with levobupivacaine after the conclusion of surgery
  Interventions: Procedure: Local wound infiltration

INTERVENTIONS:
Procedure: Superficial cervical plexus block — Patients will receive bilateral superficial cervical plexus block
  Arms: Superficial cervical plexus block
Procedure: Local wound infiltration — Patients will receive local wound infiltration
  Arms: Local wound infiltration

SUMMARY:
Tracheal resection and reconstruction (TRR) is the treatment of choice for most patients with tracheal stenosis or tracheal tumors .The postintubation tracheal stenosis is the common indication for (TRR).The immediate postoperative period can be anxiety provoking for some reasons such as requirement to maintain a flexed neck, oxygen mask, and surgical pain which inadequately treated.

Bilateral superficial cervical plexus block (BSCPB) is a popular regional anesthesia technique for its feasibility and efficacy. The use of regional anesthesia in combination with general anesthesia may lighten the level of general anesthesia required , provide prolonged postoperative analgesia and reduce the requirements for opioid analgesics

Local anesthetic infiltration into the surgical incision can relieve pain at the wound site after surgery, as part of multimodal analgesic approach.

Levobupivacaine, is "S"-enantiomer of bupivacaine, has strongly emerged as a safer alternative for regional anesthesia than bupivacaine . Levobupivacaine has been found to be equally efficacious as bupivacaine, but with a superior pharmacokinetic profile. Clinically, levobupivacaine has been observed to be well tolerated in regional anesthesia techniques both after bolus administration and continuous post-operative infusion.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the intra- and postoperative efficacy of local wound infiltration versus bilateral superficial cervical plexus block with levobupivacaine for upper tracheal resection and reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class status I or II
* Undergoing elective upper tracheal resection and reconstruction surgery

Exclusion Criteria:

* Age less than18 years
* Patients with preoperative medication included opioid
* History of allergy to the drugs used
* Coagulation disorders
* Pregnancy
* Patient refusal
* Local sepsis
* Inability to understand the study protocol or pain scale.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Estimated); Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score | For 24 hours after surgery
  Postoperative pain scores will be assessed using postoperative visual analogue score

SECONDARY OUTCOMES:
Systolic blood pressure | For 4 hours after start of surgery
Diastolic blood pressure | For 4 hours after start of surgery
Heart rate | For 4 hours after start of surgery
Peripheral oxygen saturation | For 4 hours after start of surgery
End-tidal Carbon dioxide tension | For 4 hours after start of surgery
Bispectral index | For 4 hours after start of surgery
Duration of analgesia | For 24 hours after surgery
  It is defined as time taken for first analgesic request of analgesia from extubation
Cumulative analgesic consumption | For 24 hours after surgery
  total analgesics used for 24 hrs after surgery
Cortisol serum | before induction ,one hour after start of surgery and one hour after end of surgery
  Plasma cortisol assay

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa M Elbendary, MD, Study Chair — Department of Anaesthesia, Surgical Intensive Care and Pain Medicine, College of Medicine, Mansoura University, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: Undecided